CLINICAL TRIAL: NCT07090538
Title: A Single-arm Exploratory Trial of GSL Synthetase Inhibitor Plus Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) and/ or Immune Checkpoint Inhibitor in Advanced/Metastatic Neuroblastoma.
Brief Title: GSL Synthetase Inhibitor Plus GM-CSF and/ or Immune Checkpoint Inhibitor in Previously Treated High-Risk Neuroblastoma.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-ELI-721
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: GSL synthetase inhibitor; GM-SCF
MeSH Terms: conditions — Neuroblastoma | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GM-CSF + Eliglustat (Experimental): Eliglustat 42mg will be administered twice daily in patients in the first 14 days and the following every other week until 24 weeks. For patients who still benefit from the trial, eliglustat 84mg will be administered twice daily every other week to 96 weeks.
  Prior to the initiation of Eliglustat, GM-CSF was administered for a period of five days at a dose of 250 µg/m2/day. Subsequent to this, GM-CSF is administered at a dosage of 500 µg/m2/day on Days 1-5.
  Interventions: Drug: Eliglustat

INTERVENTIONS:
Drug: Eliglustat — Drug: GM-CSF + Eliglustat Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) and GSL Synthetase Inhibitor
  Other Names: Cerdelga

SUMMARY:
This exploratory clinical study will evaluate the efficacy and feasibility of combining a GSL synthase inhibitor with a granulocyte-macrophage colony stimulating factor (GM-CSF) in patients with advanced or metastatic neuroblastoma. Six to eight eligible patients are expected to be treated in this clinical trial: 1) Assessing the anti-tumour effects of GSL synthase inhibitors in combination with immune checkpoint inhibitors and/or GM-CSF; 2) To assess immunological or clinical predictive biomarkers of efficacy and toxicity; and 3) Detecting changes in the tumour microenvironment (TME) and the dynamics of peripheral blood immune cells after treatment with a GSL synthase inhibitor combined with GM-CSF.

DETAILED DESCRIPTION:
Neuroblastoma is the most common extracranial solid tumour in infants and children. It is also known as an immunocold tumour due to the poor infiltration of immune cells in the tumour microenvironment. Tumour-associated macrophages and myeloid-derived suppressor cells account for a significant proportion of neuroblastoma cases and predominantly exert a pro-tumourigenic effect due to the tumour-suppressive microenvironment. Anti-phagocytic signals expressed by tumour cells, such as CD47, inhibit the direct cytophagy of macrophages. Patients in the high-risk group are less immunogenic and therefore less responsive to immune-checkpoint inhibitor (ICI) monotherapy than those in the low- and intermediate-risk groups. A combination of approaches may therefore be required for the immunotherapy of neuroblastoma.

Aberrant expression of glycosphingolipid (GSL) synthase is a fundamental feature of most tumours and tumour microenvironments. Neurological tumours, including neuroblastoma, have been observed to exhibit elevated levels of acidic glycosphingolipids on their surfaces. A number of studies have indicated that there is an increase in the expression of GSL synthase in tumours that are resistant to chemotherapy. Eliglustat, an oral GlcCer synthase inhibitor, has been approved for the treatment of Gaucher disease type 1. Researchers have demonstrated the excellent safety and efficacy of Eliglustat in combination with immune checkpoint inhibitors for treating advanced/metastatic solid tumours and relapsed/refractory haematological malignancies.

For these reasons, an exploratory clinical study was designed to observe the efficacy and feasibility of GSL synthase inhibitors in combination with GM-CSF in the treatment of patients with advanced/metastatic neuroblastoma. The objective of this study was to provide a high level of evidence-based rationale for the combination treatment regimen in these patients. The investigators will administer a combination of Eliglustat and GM-CSF to six patients diagnosed with advanced or metastatic NB. The primary objective of this study is to assess the efficacy and feasibility of Eliglustat in combination with GM-CSF in the treatment of neuroblastoma. The secondary objectives are to assess immunological or clinically predictive biomarkers of efficacy and toxicity, alterations in the tumour microenvironment, and changes in the dynamics of immune cells in the peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Neuroblastoma must be documented at the point of diagnosis, which is defined as one of the following: histopathology of a biopsy of a solid tumour; bone marrow aspirate or biopsy suggestive of neuroblastoma with elevated blood or urine catecholamine metabolite levels.
2. The participant is at least 6years old at time of enrollment.
3. At least one measurable lesion at baseline according to RECIST version 1.1.
4. Have adequate organ function as assessed by the laboratory required by protocol, which should be confirmed within 2 weeks prior to the first dose of study drugs.
5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity.
6. Eastern Cooperative Oncology Group (ECOG) performance status score≤2 and Estimated life expectancy of more than 3 months.
7. Patient(and/ or their parent/ legal guardian) is willing to participate and able to provide signed informed consent.

Exclusion Criteria:

1. Any systemic anti-cancer therapy, including chemotherapy or immunotherapy, within 3 weeks before 1st dose of GM-CSF
2. Existing major organ dysfunction > Grade 2, with the exception of hearing loss, hematological status, kidney and liver function
3. Active life-threatening infection
4. History of allergy or intolerance to study drug components.
5. The participant is CYP2D6 ultra-rapid metabolizer.
6. The participant is known to be allergy to Eliglustat.
7. The participant use drugs that will strongly inhibit CYP2D6 or CYP3A activity.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 120 days after the last dose of study drugs
  Objective response rate includes complete response and partial response defined by investigators according to RECIST 1.1or iRECIST criteria.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 2 years
  Time from the date of first administration of the study drug to disease progression or death from any cause (any earliest date).
Overall Survival (OS) | Up to 2 years
  Time from the date of first administration of the study drug to the date of death.

OTHER OUTCOMES:
Immunological response (cytokines, lymphocyte phenotype) | Up to 120 days after the last dose of study drugs
  Following the administration of treatment, alterations in the concentrations of cytokines (primarily nitric oxide synthase (iNOS), interleukin-1 (IL-1), interleukin-6 (IL-6), and tumour necrosis factor alpha (TNFα)) in picograms per millilitre (pg/mL)) will be evaluated in both the tumour bed and peripheral blood. Additionally, shifts in macrophage phenotypes (mainly encompassing the number and percentage of M1 and M2 cells) will be analysed using quantitative polymerase chain reaction (qPCR) and flow cytometry.
Biomarkers predictive of response and toxicity | Up to 120 days after the last dose of study drugs
  Biomarkers from tumor cells, macrophages and tumor microenvironment will be assessed for their potential in predicting clinical response and toxicity.All participants with treatment-related adverse events (AE) as assessed by National Cancer Institute Common Terminology Criteria for Adverse Event, Version 5.0(CTC AE 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (2):
- China (2):
  - Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing
  - Department of Pediatrics, The First Medical Center, Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes